CLINICAL TRIAL: NCT02903589
Title: Knowledge Attitudes, Beliefs, and Practices Regarding HIV in Populations Living on the Maroni River
Acronym: CAPMARONI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: CAPMaroni
Record Dates: First submitted 2016-09-06; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: HIV
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: observational

SUMMARY:
The HIV epidemic flared from 0 to over 1% prevalence in a decade on the Maroni river which lies between French Guiana and Surinameaim of the study is to determine the knowledge, attitudes, behaviours, and practices on HIV in the population living along the French bank of the Maroni border. Descriptive statistics are computed from the tabulation of answers to a structured questionnaire. Multivariate logistic models were computed to determine predictors of key outcomes. These data will help taylor prevention intervention in this very particular area.

ELIGIBILITY:
Inclusion Criteria:

* adult living on the maroni river

Exclusion Criteria:

* refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: general adult population living on the French bank of the maroni river
Sampling Method: Non-Probability Sample
Enrollment: 836 (Actual)
Dates: Start 2012-01; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
knowledge attitudes, beliefs, and practices regarding HIV and sexually transmitted diseases | when the interview was conducted
  a structured questionnaire was used.. it was administered face to face with usually 5 possible responses. Scores were established using similar questions exploring related areas of HIV.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Cayenne, Cayenne, French Guiana, France